CLINICAL TRIAL: NCT03893409
Title: A Observational Study in Chinese Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: GIRH Chronic Obstructive Pulmonary Disease Observational Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: zili zhang (Other)
Responsible Party: Sponsor-Investigator, zili zhang, Guangzhou Medical University, The First Affiliated Hospital of Guangzhou Medical University
Organization: The First Affiliated Hospital of Guangzhou Medical University (Other)
Other Study IDs: Respiratory disease of GIRH
Record Dates: First submitted 2019-03-26; First posted 2019-03-28 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pulmonary function
- biological sample detection outcome

INTERVENTIONS:
Other:  — this is a observation study, no any intervention in patients

SUMMARY:
The purpose of this study is to establish the large COPD cohort and biological database in China, aiming for precision medicine to optimize diagnosis and treatment choices.

ELIGIBILITY:
Inclusion Criteria:

-Aged 40-70 years COPD group: baseline post-bronchodilator FEV1/FVC < 0.7 Signed informed consent obtained prior to participations with the ability to comply with protocol and be available for study visits over 5 years

Exclusion Criteria:

* Acute exacerbation in the past 3 months Having other respiratory diseases with massive lung tissue destruction such as severe bronchiectasis and tuberculosis, etc The usual criteria of serious uncontrolled diseases thoracic or abdominal surgery in the last 3 months eye surgery in the last three months retinal detachment myocardial infarction in the last 3 months admission to hospital for any cardiac condition in the last month heart rate over 120 beats per minute antibacterial chemotherapy for tuberculosis pregnant or breast feeding

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a observational prospective longitudinal cohort study to to establish the large COPD cohort and biological database in China, including COPD subjects( n= 5000) and healthy subjects (n= 5000). Sites Investigators will be respiratory physicians working in the respiratory department of our sites, which must be tier 2 or tier 3 hospitals in China, with the equipment and ability to conduct pulmonary function test, HRCT. Patients must meet all the inclusion criteria and none of the exclusion criteria. No additional investigational drugs will be applied to the patients. Statistical analysis will be conducted by epidemiology & statistics work group from Chinese Academy of Sciences, using SAS and R software. Paper-based questionnaire administration will also be used. Questionnaire variables will be checked before data entry. During the study, PI will be in charge of the monitoring of the whole procedure.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2018-08-10 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
difference of FEV1 at 12 months from baseline | at 12 months
  difference of FEV1 at 12 months from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes